CLINICAL TRIAL: NCT06378476
Title: Using Community Health Workers and Trauma-Informed Care Training for Clinicians to Improve Kidney Disease Outcomes in a Diverse Urban Community
Brief Title: Supportive Understanding and Patient-centered Partnership for Optimizing Renal Treatment
Acronym: SUPPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Judith Long, MD, Sol Katz Professor of Medicine, University of Pennsylvania Perelman School of Medicine; Chief, Division of General Internal Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 855188
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Diseases; Racism, Systemic; Trauma, Psychological
MeSH Terms: conditions — Renal Insufficiency, Chronic; Systemic Racism; Psychological Trauma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research coordinators collecting baseline and outcomes data from participants will be blinded to arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHW + TIC (Experimental): Patients in this arm will receive 6 months of support from a community health worker as well as primary care from a clinic where clinicians and staff have undergone trauma-informed care training.
  Interventions: Behavioral: IMPaCT Community Health Worker Program; Other: Trauma-Informed Care Training
- TIC only (Experimental): Patients in this arm will receive primary care from a clinic where clinicians and staff have undergone trauma-informed care training.
  Interventions: Other: Trauma-Informed Care Training
- Usual Care (No Intervention): Patients in this arm will receive usual care.

INTERVENTIONS:
Behavioral: IMPaCT Community Health Worker Program — The IMPaCT intervention consists of three stages: goal-setting, tailored support, and connection with long-term support. CHWs first seek to understand the patient's individual circumstances, life histories, and priorities by using a semi-structured interview guide inquiring about social and behavioral determinants of health. CHWs will then partner with patients to create customized action plans based on patient needs.
  Arms: CHW + TIC
Other: Trauma-Informed Care Training — Primary care providers and staff at two General Internal Medicine clinics will receive training in providing supportive care to patients who have experienced trauma. The trainings are all action focused and include a review of racism in medicine, understanding intergenerational trauma and its impact on care, naming and mitigating barriers to health equity, and the basics of motivational interviewing
  Arms: CHW + TIC; TIC only

SUMMARY:
Black and Hispanic people face higher risks of chronic kidney disease (CKD) but have unequal access to the highest-quality kidney care. Black adults with CKD face 1.5 times higher hospitalization risks than non-Black adults with CKD. Once reaching end stage kidney disease (ESKD), Black patients are half as likely to receive a transplant and are often excluded from home dialysis. Structural racism creates complex barriers to optimal CKD care, providing an explanation for these findings. The Penn Medicine IMPaCT Community Health Worker (CHW) program is a rigorously tested approach to employ people from local communities to dismantle structural racism within health care systems and improve outcomes for marginalized patients. This trial will innovate by training CHWs to focus specifically on CKD care for minoritized people. The investigators will also train primary care clinicians caring for CKD patients on how to provide trauma-informed care (TIC). The first aim is to determine the feasibility, acceptability, and reach of a clinic-level TIC training to address the needs and concerns of Black and other minoritized patients. The second aim will be to conduct a three arm trial comparing individuals in usual care to individuals randomized to either our tailored CHW intervention in conjunction with clinic-level TIC training or to clinic-level TIC intervention only. The investigators will examine whether patients in the intervention arms have greater improvements in quality of life (primary). The investigators will also explore the impact of the interventions on patient activation, hospitalizations, and ESKD treatment preferences.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stage 4 or 5
* Patient at participating general internal medicine or family medicine clinic
* Medicaid-eligible or uninsured
* Reside in high poverty Philadelphia zip code

Exclusion Criteria:

* No history of kidney transplant
* Not receiving any form of dialysis
* Not previously enrolled with a community health worker in the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Kidney Disease Quality of Life Instrument (KDQOL) | 6 months
  KDQOL-36 is a short form that includes a generic score (the 12-Item Short Form Health Survey (SF-12), which includes the SF-12 Physical and Mental Component Summaries [SF-12 PCS and MCS]) and three CKD-specific subscales: 1) burden of kidney disease, 2) symptoms/problems of kidney disease, and 3) effects of kidney disease. Each of the KDQOL-36 kidney-targeted scales are scored by transforming all items linearly to a 0-100 possible range and averaging the items in the scale. On the KDQOL-36, higher scores indicate better health-related quality of life.

SECONDARY OUTCOMES:
Patient Activation Measure | 6 months
  The 10-item self-reported Patient Activation Measure (PAM) assesses patient knowledge, skill, and confidence for self-management of health conditions. The PAM provides an individual 'activation' score on a 0-100 point scale. Higher scores indicate greater activation.
All-Cause Hospitalizations | 6 months
  The investigators will ascertain hospitalizations for 6 months after randomization via: a) participant report (with confirmation from a secondary source), b) electronic health records, and c) the Pennsylvania HealthCare Cost Containment Council (PHC4), which captures every hospitalization in the state and has diagnostic codes for hospitalization cause.
Patient preferences for end-stage renal disease treatment | 6 months
  To measure treatment preferences, we will ask patients what treatment they would select today if they needed renal replacement therapy (RRT) now - transplant, in-center dialysis, home dialysis, or palliative care.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States